CLINICAL TRIAL: NCT03300167
Title: Study of the Vascular Response to Percutaneous Coronary Intervention in Patients With Non-ST-elevation Acute Coronary Syndromes Using Intravascular Blood Sampling
Acronym: IN HEART
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Delivery of equipment. PI not had any further interaction with the company so closed study.
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STH19267
Record Dates: First submitted 2017-06-13; First posted 2017-10-03 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-11

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CE-marked coronary artery catheter (Experimental): use of a novel CE-marked coronary artery catheter to obtain spatially-separated intravascular samples for laboratory measurement.
  Interventions: Device: The Liquid Biopsy System

INTERVENTIONS:
Device: The Liquid Biopsy System — The Liquid Biopsy System is a single use percutaneously-delivered coronary blood sampling device designed to collect blood samples from within a target coronary artery so that the blood can be analysed.

SUMMARY:
This interventional study is using the PlaqueTec LBS will enrol participants already undergoing coronary angiography as a component of their standard care for NSTE-ACS. The study will involve no change to medication or overall treatment strategy, but will involve an additional procedure: use of a novel CE-marked coronary artery catheter to obtain spatially-separated intravascular samples for laboratory measurement. As a safety objective and as a component of the required post-marketing surveillance, OCT will be performed before and after deployment of the LBS, and patients will be followed up for a significant period of time by the investigator's post-procedure.

Individual participants will not gain directly from taking part in the study, other than having access to more prolonged follow up than is standard. However, new insights will be gained into the microenvironment surrounding a ruptured plaque in NSTE-ACS, which has the potential to benefit patients with CAD in the future through greater understanding of the effects of current therapy, development of new treatment strategies and methods of assessing the efficacy of those treatment strategies.

Use of the LBS and the associated OCT examinations will require additional angiographic screening and therefore lead to greater exposure to radiation and higher contrast load. This will be closely monitored as per Trust policies in line with IRMER and local radiological guidelines. Patients at particular risk of developing complications from increased exposure to radiation and contrast (eg. those who are pregnant and those with abnormal baseline renal function) will not be included in order to minimise adverse effects.

DETAILED DESCRIPTION:
This clinical protocol will be subject to peer review according to standard local procedures, including independent scientific review by the Scientific Advisory Board of the Clinical Research Facility, Sheffield Teaching Hospitals NHS Foundation Trust; the Clinical Research Office, Sheffield Teaching Hospitals NHS Foundation Trust; and the Research Ethics Committee. The study will be a single-centre study including use of a CE-marked medical device to obtain samples, conducted at Cardiology and Cardiothoracic Surgery Directorate, Northern General Hospital, Sheffield Teaching Hospitals NHS Foundation Trust.

Patients with a diagnosis of NSTE-ACS, receiving DAPT with a combination of aspirin and ticagrelor or prasugrel, and listed either for coronary angiography with the intention of proceeding to PCI or for PCI following coronary angiography at a referring hospital, will be approached and their informed consent sought for this study. 18 patients found to have culprit significant proximal epicardial coronary artery stenosis suitable for PCI, meeting all the inclusion and exclusion criteria, will proceed to have platelet function testing and LBS measurements. Blood will be taken from the arterial sheath or guide catheter and baseline platelet function testing will be performed (VerifyNow P2Y12 assay; light transmittance aggregometry with ADP and arachidonic acid as agonists; and serum thromboxane B2 assay). Balloon predilatation prior to stent deployment will be a mandatory requirement for the study. Following balloon predilatation, the LBS will be deployed across the treated lesion and blood sampling will be performed proximal and distal to the lesion at approximately 5 minutes after predilatation. The following assays will be performed on the sampled blood:

1. Plasma levels of soluble markers of thrombosis and inflammation including prothrombin fragments 1 and 2, fibrinopeptide A, soluble P-selectin and thromboxane B2.
2. Platelet surface P-selectin expression
3. Leukocyte surface CD11b expression Blood taken prior to PCI will also be sent to the local laboratory for measurement of the cardiac-specific marker high-sensitivity troponin T and a further venous blood sample will be collected at 6 hours after PCI to measure any rise in troponin in order to correlate this with thrombin generation. A rise of 5 times the upper limit of normal of troponin following PCI in the context of chest pain or diagnostic ECG changes will be used to define peri-procedural myocardial infarction per the Universal Definition of Myocardial Infarction (Thygesen, Alpert et al. 2012).

OCT of the culprit lesion, as well as the coronary artery proximal and distal to this, will be performed before and after the deployment of the LBS to assess any topographical changes to the vessel wall caused by the LBS and provide information on target lesion morphology.

Clinical outcomes will be reviewed and AEs (including MACE) will be recorded at 6 hours, 30 days and 6 months after the procedure. At the 6-hour visit, patients will be assessed by a medically-qualified investigator and have a blood sample collected for troponin T level and ECG performed. At the 30-day visit, patients will receive a full clinical assessment by a medically-qualified investigator, have DAPT compliance assessed, be asked about angina intensity, have any MACE or other AEs recorded and have an ECG. A telephone contact will be made at 6 months after PCI to assess any MACE or other AEs, angina intensity and DAPT compliance.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Admitted to hospital with non-ST-elevation ACS and plan for either coronary angiography with a view to PCI if appropriate or PCI following coronary angiography at a referring hospital
* Current treatment with aspirin and ticagrelor or, if ticagrelor is not tolerated, prasugrel (DAPT)
* Ability to give informed consent

Exclusion Criteria:

* Treatment with antiplatelet medication apart from aspirin, ticagrelor, prasugrel or clopidogrel in the last 10 days (e.g. dipyridamole, abciximab, tirofiban).
* Planned use of a glycoprotein IIb/IIIa antagonist for the PCI procedure.
* Patients with haemodynamic instability, shock or angiographic evidence of intracoronary thrombus.
* Current use of an oral anticoagulant (e.g. warfarin, dabigatran, rivaroxaban, apixaban).
* Clinically significant liver disease.
* Contraindication or allergy to unfractionated heparin.
* Receiving immunosuppressant medication (eg. cyclosporin, tacrolimus, mycophenolate, azathioprine).
* Administration of doses of low molecular weight heparin or fondaparinux in the 12 hours preceding PCI.
* Known severe left ventricular dysfunction (ejection fraction <30%).
* Culprit lesion in left main coronary artery.
* Women of childbearing potential unless pregnancy has been excluded during the index hospital admission.
* Known serum creatinine above upper limit of local reference range.
* Subjects with known active chronic inflammatory disease, e.g. systemic lupus erythematosus, rheumatoid arthritis, seropositive arthropathies and known seropositivity to HIV, Hepatitis B or Hepatitis C.
* Severely diseased, excessively tortuous or calcified coronary vessels that increase the risk of snaring the LBS.
* Culprit lesion in a coronary vessel with a reference diameter of less than 2.5 mm.
* Need to cross a region of coronary vessel that contains a stent.
* Evidence of ongoing sepsis.
* Receiving a non-steroidal anti-inflammatory drug (NSAID) apart from aspirin, including selective COX2 inhibitors ('coxibs') and including regular or intermittent/as required use.
* Receiving a strong inhibitor of CYP3A4 (eg, ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin [but not erythromycin or azithromycin], nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atanazavir, or over 1 litre daily of grapefruit juice).
* Receiving simvastatin or lovastatin at doses higher than 40 mg daily.
* Receiving a CYP3A substrate with a narrow therapeutic index (e.g. cyclosporine or quinidine).
* Receiving a strong inducer of CYP3A (e.g. rifampin/rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital).
* Current or recent (within 30 days) participation in a clinical trial of a drug or device or any other clinical study that might influence the results or safety of the study.
* Any factor precluding ability to comply with follow-up.
* Any other factor judged by the investigator or treating physician to preclude enrolment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma prothrombin fragments | during the percutaneous coronary intervention procedure
  Plasma prothrombin fragments 1+2 compared within-patients between samples from distal, mid and proximal ports

SECONDARY OUTCOMES:
Fibrinopeptide A | during the percutaneous coronary intervention procedure and 6 hours later [peri-procedural MI only]
  Compared with 0-6 hour serum hsTnT rise
Soluble platelet P-selectin | during the percutaneous coronary intervention procedure and 6 hours later [peri-procedural MI only]
  Compared with 0-6 hour serum hsTnT rise
TXB2 | during the percutaneous coronary intervention procedure and 6 hours later [peri-procedural MI only]
  Compared with 0-6 hour serum hsTnT rise
platelet surface P-selectin expression | during the percutaneous coronary intervention procedure and 6 hours later [peri-procedural MI only]
  Compared with 0-6 hour serum hsTnT rise
Leukocyte surface CD11b expression | during the percutaneous coronary intervention procedure and 6 hours later [peri-procedural MI only]
  Compared with 0-6 hour serum hsTnT rise

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kavanagh TG, Griffiths NJ, Todd I. Psoas abscess and Crohn's disease. J R Soc Med. 1979 Aug;72(8):612-3. doi: 10.1177/014107687907200813. No abstract available. PMID 552561
- [Background] Caine ED, Polinsky RJ. Haloperidol-induced dysphoria in patients with Tourette syndrome. Am J Psychiatry. 1979 Sep;136(9):1216-7. doi: 10.1176/ajp.136.9.1216. No abstract available. PMID 289300
- [Background] Timmermans PJ, Vossen JM. Prey catching in the archer fish: does the fish use a learned correction for refraction? Behav Processes. 2000 Oct 26;52(1):21-34. doi: 10.1016/s0376-6357(00)00107-8. PMID 11011106
- [Background] Suzuki N, Kato M, Dohmori R. [Synthesis of antimicrobial agents. II. Synthesis of 1,8-naphthyridine derivatives and their activities against Trichomonas vaginalis (author's transl)]. Yakugaku Zasshi. 1979 Feb;99(2):155-64. doi: 10.1248/yakushi1947.99.2_155. No abstract available. Japanese. PMID 312317
- [Background] Lai Y, Xu DP. [Study on the chemical structure from the roots of Actinidia deliciosa]. Zhong Yao Cai. 2007 Feb;30(2):166-8. Chinese. PMID 17571763
- [Background] [Animal husbandry (the main trends)]. Veterinariia. 1977 Jun;(6):LL'*23. No abstract available. Russian. PMID 929940
- [Background] May A. The Confidential Enquiries into Maternal Deaths 1997-1999: what can we learn? Int J Obstet Anesth. 2002 Jul;11(3):153-5. doi: 10.1054/ijoa.2002.0957. No abstract available. PMID 15321539
- [Background] Falgoust DL. Hospital security over the years: keeping up with the changes. J Healthc Prot Manage. 2002 Summer;18(2):115-22. PMID 12371242
- [Background] da Costa MC. [Correlation between serum DDT levels and the diphtheria antibody titer in girls]. Rev Saude Publica. 1979 Mar;13(1):32-42. doi: 10.1590/s0034-89101979000100005. No abstract available. Portuguese. PMID 223229
- [Background] Courtney LD. Respiratory distress syndrome. Br Med J. 1977 Mar 5;1(6061):639. doi: 10.1136/bmj.1.6061.639-a. No abstract available. PMID 843850
- [Background] Farng E, Hunt SA, Rose DJ, Sherman OH. Anterior cruciate ligament radiofrequency thermal shrinkage: a short-term follow-up. Arthroscopy. 2005 Sep;21(9):1027-33. doi: 10.1016/j.arthro.2005.05.015. PMID 16171626
- [Background] Costa M, Pecci L, Pensa B, Cannella C. Hydrogen peroxide involvement in the rhodanese inactivation by dithiothreitol. Biochem Biophys Res Commun. 1977 Sep 23;78(2):596-603. doi: 10.1016/0006-291x(77)90221-2. No abstract available. PMID 410413
- [Background] Mertz D, Johnstone J, Loeb M. Does duration of perioperative antibiotic prophylaxis matter in cardiac surgery? A systematic review and meta-analysis. Ann Surg. 2011 Jul;254(1):48-54. doi: 10.1097/SLA.0b013e318214b7e4. PMID 21412147
- [Background] Zagury D, Chaouat G, Morgan DA, Voisin GA. [Identification of cytotoxic cells responsible for lysis of target cells pretreated with concanavalin A in spleen populations of pregnant mice with suppressive activity]. C R Seances Acad Sci D. 1979 May 7;288(17):1343-6. French. PMID 113118
- [Background] Donnelly N, Hadwin JA, Cave K, Stevenage S. Perceptual dominance of oriented faces mirrors the distribution of orientation tunings in inferotemporal neurons. Brain Res Cogn Brain Res. 2003 Oct;17(3):771-80. doi: 10.1016/s0926-6410(03)00201-5. PMID 14561462
- [Background] Niederer RO, Zappulla DC. Refined secondary-structure models of the core of yeast and human telomerase RNAs directed by SHAPE. RNA. 2015 Feb;21(2):254-61. doi: 10.1261/rna.048959.114. Epub 2014 Dec 15. PMID 25512567
- [Background] Megla GK. [A new blood gas analyzer Corning model 175]. Med Lab (Stuttg). 1976 Jan;29(1):12-22. No abstract available. German. PMID 8691
- [Background] Pongrakhananon V, Luanpitpong S, Stueckle TA, Wang L, Nimmannit U, Rojanasakul Y. Carbon nanotubes induce apoptosis resistance of human lung epithelial cells through FLICE-inhibitory protein. Toxicol Sci. 2015 Feb;143(2):499-511. doi: 10.1093/toxsci/kfu251. Epub 2014 Nov 19. PMID 25412619
- [Background] Statement on flexible patterns of nursing education. ANA Publ. 1978;(NE-3):i-iv, 1-13. No abstract available. PMID 249257